CLINICAL TRIAL: NCT02578095
Title: A Phase II, Randomized, Double-Blind, Parallel Group, Placebo- Controlled, Multi-Center Study to Explore the Efficacy, Safety and Tolerability of VK5211 in Subjects With Acute Hip Fracture
Brief Title: Acute Hip Fracture Study in Patients 65 Years or Greater
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viking Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VK5211-201
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo QD
  Interventions: Drug: Placebo
- VK5211- 0.5mg (Experimental): 0.5mgQD
  Interventions: Drug: VK5211
- VK5211- 1.0mg (Experimental): 1.0mg QD
  Interventions: Drug: VK5211
- VK5211- 2.0mg (Experimental): 2.0mg QD
  Interventions: Drug: VK5211

INTERVENTIONS:
Drug: VK5211 — Capsule
  Arms: VK5211- 0.5mg; VK5211- 1.0mg; VK5211- 2.0mg
Drug: Placebo — Capsule
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, parallel group, placebo-controlled, multicenter study to investigate the safety, tolerability, and efficacy of VK5211 after 12 weeks of treatment.

Males and females ≥65 years old who are ambulatory and recovering from a hip fracture will be eligible for participation 3-7 weeks post-injury.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥65 years old who are recovering from a hip fracture (occurring 3-7 weeks prior) with no residual surgical issues will be eligible for participation.

Exclusion Criteria:

* Pathological fracture (e.g. fracture due to Paget's disease of bone, malignancy, etc.). Fracture due to postmenopausal osteoporosis is not considered pathological for this trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Mancini, Study Director — Viking Therapeutics, Inc.
Locations (21):
- United States (7):
  - Duurga Clinical Service, Yorba Linda, California
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Infinite Clinical Research, Doral, Florida
  - Shrock Orthopedic Research, LLC, Fort Lauderdale, Florida
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Orthopaedic Association of Michigan, Grand Rapids, Michigan
  - University of Wisconsin Osteoporosis Clinical Research Program, Madison, Wisconsin
- Hungary (6):
  - Szent János Kórház és Észak budai Egyesített Kórházak Traumatológiai és Kézsebészeti Osztály, Budapest
  - MH Egészségügyi Központ Baleseti Sebészeti Osztály, Budapest
  - Szent Margit Kórház, Mozgásszervi Rehabilitációs Osztály, Budapest
  - Petz Aladár Megyei Oktató Kórház Mozgásszervi Rehabilitációs Osztály, Győr
  - Jósa András Oktató Kórház Traumatológiai és Kézsebészeti Osztály, Nyíregyháza
  - SZTE ÁOK Traumatológiai Klinika, Szeged
- Romania (3):
  - Spitalul Clinic de Urgenta Bucuresti ("Floreasca"), Bucharest
  - Spitalul Universitar de Urgenţă, Bucharest
  - Spitalul Clinic Judeţean de Urgenţe, Sfȃntul Spiridon, Iași
- Serbia (5):
  - Institut za Ortopedsko-hirurške bolesti Banjica, Belgrade
  - Klinički Centar Srbije, Belgrade
  - Hospital Center "Bezanijska kosa" Department for Orthopedic Surgery and Traumatology, Belgrade
  - Clinical Center Kragujevac Department for Orthopedics and Traumatology, Kragujevac
  - Clinical Centre of Vojvodina Department for Orthopedic Surgery and Traumatology, Novi Sad

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | VK5211- 0.5mg | VK5211- 1.0mg | VK5211- 2.0mg
Started | 28 | 29 | 26 | 25
Completed | 19 | 22 | 17 | 17
Not Completed | 9 | 7 | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | VK5211- 0.5mg | VK5211- 1.0mg | VK5211- 2.0mg | Total
Number analyzed (Participants) | 28 | 29 | 26 | 25 | 108
Age, Continuous [Median (Full Range); unit: Years] | 76 [64 to 91.7] | 78 [65 to 86] | 78.5 [65 to 94] | 78 [65 to 93.7] | 78 [64 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 22 | 19 | 83
  Male | 9 | 6 | 4 | 6 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 29 | 24 | 25 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 27 | 0 | 0 | 0 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy in Hip Fracture Patients Confirmed by DXA Scan.
Description: Efficacy of VK5211 after 12 weeks of treatment by mean placebo-corrected percentage change in total body less head (TBLH) lean body mass assessed by whole body dual-energy x-ray absorptiometry scan (DXA) scan.
Time Frame: Baseline and Week12
Population: The ITT population was the primary analysis population for assessing efficacy.
Measure: Least Squares Mean (95% Confidence Interval); unit: PBO adjusted percent change
Arm/Group | Placebo | VK5211- 0.5mg | VK5211- 1.0mg | VK5211- 2.0mg
Number analyzed (Participants) | 20 | 27 | 17 | 15
PBO adjusted percent change | 0 [0 to 0] | 4.75 [1.70 to 7.80] | 7.15 [3.76 to 10.54] | 9.08 [5.55 to 12.60]
Statistical Analysis 1: Comparison: Placebo vs VK5211- 0.5mg; Test type: Superiority; p = 0.0032, ANCOVA; Mean Difference (Final Values) = 4.75, 95% CI 2-sided [1.70 to 7.80]
Statistical Analysis 2: Comparison: Placebo vs VK5211- 1.0mg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 7.15, 95% CI 2-sided [3.76 to 10.54]
Statistical Analysis 3: Comparison: Placebo vs VK5211- 2.0mg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 9.08, 95% CI 2-sided [5.55 to 12.60]

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Placebo | VK5211- 0.5mg | VK5211- 1.0mg | VK5211- 2.0mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 4/28 | 2/29 | 3/26 | 5/25
Other Adverse Events (participants affected / at risk) | 10/28 | 11/29 | 8/26 | 16/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | VK5211- 0.5mg (N=29) | VK5211- 1.0mg (N=26) | VK5211- 2.0mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroxine Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | VK5211- 0.5mg (N=29) | VK5211- 1.0mg (N=26) | VK5211- 2.0mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Valve Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyrodism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increase (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate Aminotransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Alkaline Phosphatase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
International Normalised Ration Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver Function Test Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroxine Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal Loss of Weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pubic Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral Ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Field Defect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterovaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Circulatory Collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-12-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT02578095/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT02578095/SAP_003.pdf